CLINICAL TRIAL: NCT05650372
Title: Comparison Of The Efficiency Of High Intensity And Low Intensity Resistive Exercises In Patient With Upper Extremity Lymphedema
Brief Title: High Intensity vs Low Intensity Resistive Exercise In Patient With Upper Extremity Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc. Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-KAEK-64-22-09
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lymphedema
Keywords: Lymphedema; Resistive Exercises
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind study
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blind to the randomization and the investigator will be blind to the outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity resistive exercise group (Experimental): Participants of this group will be applied manual lymphatic drainage and compression bandaging and they will exercise for 25 minutes, three sets of each exercise at 80% intensity of 1 max repetition.
  Interventions: Other: High intensity resistive exercise
- Low intensity resistive exercise group (Active Comparator): Participants in this group will be applied manual lymphatic drainage and compression bandaging and they will exercise for 25 minutes, three sets of each exercise at 30% intensity of 1 max repetition.
  Interventions: Other: Low intensity resistive exercise

INTERVENTIONS:
Other: High intensity resistive exercise — Participants of this group will be applied manual lymphatic drainage and compression bandaging every day of the week, and they will exercise for 25 minutes, three sets of each exercise at 80% intensity of 1 max repetition, 2 days of the week. Exercise training consist of warm-up and cool-down (10-15 repetitions of range of motion and 10 minutes of active stretching exercises) and resistive exercises.Each of the experimental sessions involved resistance exercises targeting all the major muscle groups in the upper body. Specifically, the exercises included the chest press, lat pull-down, bicep curl, triceps extension, lateral raise, and wrist curl.
  Arms: High intensity resistive exercise group
Other: Low intensity resistive exercise — participants in this group will be applied manual lymphatic drainage and compression bandaging every day of the week and they will exercise for 25 minutes, three sets of each exercise at 30% intensity of 1 max repetition 2 days of the week.
  Exercise training consist of warm-up and cool-down (10-15 repetitions of range of motion and 10 minutes of active stretching exercises) and resistive exercises. Each of the experimental sessions involved resistance exercises targeting all the major muscle groups in the upper body. Specifically, the exercises included the chest press, lat pull- down, bicep curl, triceps extension, lateral raise, and wrist curl.
  Arms: Low intensity resistive exercise group

SUMMARY:
Lymphedema results from impaired lymphatic transport with increased limb volume. The results of systematic reviews indicate that breast cancer survivors can perform resistance exercise training at high-enough intensities to elicit strength gains without triggering changes to lymphedema status. There is strong evidence indicating that ret produces significant gains in muscular strength without provoking breast cancer-related lymphedema. On the one hand, the literature studies say future exercise programs will have to be evaluated in detail regarding intensity, volume, duration, frequency, and exercised muscle group. The purpose of this study is to examine the impact of upper body resistance exercise on the arm circumference, grip strength, pain, musculoskeletal disorders of the upper limbs, self-reported lymphedema symptoms, pinch strength, lymphedema functioning, disability, and health questionnaire/lymph-ıcf patient with upper extremity lymphedema and to compare these effects between resistance exercise involving high and low loads (heavier vs lighter weights).

DETAILED DESCRIPTION:
Lymphedema results from impaired lymphatic transport with increased limb volume.

Lymphedema is divided into primary and secondary forms. Secondary lymphedema is likely to occur after the surgical removal of lymph nodes or in conjunction with radiotherapy. Secondary lymphedema is generally described as arm swelling and dysfunction. It is defined as an increase in arm circumference by more than 2 cm or as an accumulation of excessive protein-rich liquid in a part of the body where lymphatic vessels have been damaged. Erysipelas (cellulitis) is the main complication, but psychological or functional discomfort may occur throughout the course of lymphedema. The associated swelling may range from mild to disabling and is associated with feelings of distress, heaviness, and weakness in the arm, pain, and an increased risk for infection. These symptoms further impair the functional and self-care abilities of the individuals, causing significant psychological distress and reduced quality of life. Upper-limb lymphedema secondary to breast cancer treatment is the most frequent. Lymphedema management is based on complete decongestive physiotherapy (multilayer low-stretch bandage, manual lymph drainage, skincare, and exercises). The American college of sports medicine (ACSM) roundtable on exercise guidelines for cancer survivors describes that exercise during and after cancer treatment is safe and can help patients improve their physical capacity and quality of life. The ACSM guidelines indicate specific exercise programs oriented towards impairments associated with disease and medical treatment. Strength exercise does not have any adverse effects on an existing to; instead, it has beneficial effects such as improvement of strength and lower exacerbation rates. For breast cancer survivors who develop lymphedema, resistance exercise has been demonstrated to improve symptom severity, strength, endurance, and mobility of the affected limb, without exacerbating lymphedema. Recent evidence indicates that resistance exercise training can be an effective management strategy for breast cancer-related lymphedema by improving functional capacity and lymph flow through the pumping effect stimulated by muscular contraction. The results of systematic reviews indicate that breast cancer survivors can perform resistance exercise training at high-enough intensities to elicit strength gains without triggering changes to lymphedema status. There is strong evidence indicating that ret produces significant improvements in muscular strength without provoking breast cancer-related lymphedema. On the one hand, the literature studies say future exercise programs will have to be evaluated in detail regarding intensity, volume, duration, frequency, and exercised muscle group. The purpose of this study is examine the impact of upper body resistance exercise on the arm circumference, grip strength, pain, musculoskeletal disorders of the upper limbs, self-reported lymphedema symptoms, pinch strength, lymphedema functioning, disability, and health questionnaire/lymph-ıcf patient with upper extremity lymphedema and to compare these effects between resistance exercise involving high and low loads (heavier vs lighter weights).

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with lymphedema of the upper extremity at least 6 months ago by the physician
* Having stage 2 lymphedema
* Having a circumference difference of 2-8 cm at any reference point between the affected extremity and the healthy extremity
* Being between the ages of 35-60
* Volunteer to participate
* Not receiving lymphedema treatment in the last 6 months

Exclusion Criteria:

* Having stage 1 or 3 lymphedema
* Have a greater than 8 cm less than 2 cm circumference difference any reference point between the affected extremity and the healthy extremity
* Papilloma, lymphedema or elephanthiasis with hyperkeratosis
* Have acute inflammatory diseases

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Arm circumference measurement | 1 month
  Bilateral arm circumference will be measured using a measuring tape at six reference points:
  the metacarpophalangeal joint, wrist joint, 10 and 15 cm distal to the lateral epicondyle, and 10 and 15 cm proximal to the lateral epicondyle.

SECONDARY OUTCOMES:
Measure of grip strength | 1 month
  Grip strength on the affected extremity will be measured with a jamar dynamometer.
Evaluation of pain (McGill Pain Questionnaire) | 1 month
  The mcgill Pain Questionnaire is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The questionnaire is a multi-dimesional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain.
The disabilities of the arm, shoulder and hand (DASH) questionnaire | 1 month
  Assess musculoskeletal disorders of the upper limbs will be measured this questionnaire.
  The disabilities of the arm, shoulder, and hand questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms.
Lymphedema Life Impact Scale | 1 month
  Lymphedema Life Impact Scale was developed as a comprehensive,lymphedema-specific instrument to assess the effects of lymphedema on any extremity. The questionnaire is an 18-item measure of physical, psychosocial, and functional impairments caused by lymphedema.
Lymphedema Symptom Severity Scale | 1 month
  The subjective feeling of heaviness, swelling, and tension intensity will be measured using a visual analog scale.
Pinch Strength Test | 1 month
  This evaulation for measuring the maximum isometric strength of the hand and forearm muscles when doing a pinching action and pinch strength on the affected extremity will be measured with a pinch meter.
Lymphedema Functioning, Disability and Health Questionnaire | 1 month
  The Lymphedema Functioning, Disability, and Health Questionnaire is a reliable and valid questionnaire to assess impairments in function, activity limitations, and participation restrictions of patients with arm lymphedema after axillary dissection for breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akinci, PT, PhD, Study Chair — Biruni University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No